CLINICAL TRIAL: NCT04425746
Title: A Phase II, Multicentre, Double-blind, Placebo Controlled, Pilot Study to Evaluate the Safety and Efficacy of CUV1647 (Afamelanotide) as Adjunctive Therapy in Patients Undergoing Photodynamic Therapy (PDT) Utilising Porfimer Sodium
Brief Title: Afamelanotide as Adjunctive Therapy in Patients Undergoing Photodynamic Therapy (PDT) Utilising Porfimer Sodium
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clinuvel Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CUV025
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Results first posted 2021-10-01 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Patients Undergoing Photodynamic Therapy Using Porfimer Sodium
MeSH Terms: interventions — afamelanotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Afamelanotide (Experimental): Subjects visited the clinic on Day 0 (administration of afamelanotide implant and porfimer sodium), Day 2 (photodynamic therapy), and Days 20 and 90 for assessments of adverse events, concomitant medication and the results of evaluation of phototoxicity.
  Interventions: Drug: Afamelanotide
- Placebo (Placebo Comparator): Subjects visited the clinic on Day 0 (administration of placebo implant and porfimer sodium), Day 2 (photodynamic therapy), and Days 20 and 90 for assessments of adverse events, concomitant medication and the results of evaluation of phototoxicity.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Afamelanotide
  Arms: Afamelanotide
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study was to evaluate the safety and efficacy of afamelanotide (previously developed as CUV1647) as adjunctive therapy in patients undergoing photodynamic therapy using porfimer sodium.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Caucasian subjects undergoing photodynamic therapy with porfimer sodium;
* Aged greater than 18 years;
* Written informed consent prior to the performance of any study-specific procedure.

Exclusion Criteria:

* Known allergy or hypersensitivity to afamelanotide or the polymer contained in the implant;
* Non-Caucasian patients;
* Personal history of melanoma or dysplastic nevus syndrome;
* Current Bowen's disease, basal cell carcinoma, squamous cell carcinoma, or other malignant or premalignant skin lesions;
* Female who is pregnant (confirmed by positive serum β-HCG pregnancy test prior to baseline) or lactating;
* Females of child-bearing potential (pre-menopausal, not surgically sterile) not using adequate contraceptive measures (i.e. oral contraceptives, diaphragm plus spermicide, intrauterine device);
* Participation in a simultaneous clinical trial for another investigational agent or within 30 days prior to the screening visit;
* Patients unable to give informed consent;
* Patient needs for concomitant medication with potential photosensitizing effects e.g. antibiotics like tetracyclines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-08-05 (Actual); Primary Completion 2009-05-28 (Actual); Study Completion 2009-05-28 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Afamelanotide: Subjects visited the clinic on Day 0 (administration of afamelanotide implant and porfimer sodium), Day 2 (photodynamic therapy), and Days 20 and 90 for assessments of adverse events, concomitant medication, and the results of evaluation of phototoxicity.
Period: Overall Study
Arm/Group | Afamelanotide | Placebo
Started | 9 | 7
Completed | 9 | 6
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Afamelanotide | Placebo | Total
Number analyzed (Participants) | 9 | 7 | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.0 (9.3) | 72.6 (8.8) | 67.2 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 9 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: The First Day on Which Patients Are Free From Symptoms of Phototoxicity Following Phototesting
Time Frame: From Day 04 to Day 90
Population: The planned primary efficacy endpoint was the number of days for patients to be free of phototoxic reactions following phototesting. This was recorded by patients through diaries, however these diaries were not completed appropriately, thus data could not be collected. Thus, the efficacy analysis was performed using the secondary efficacy endpoint, change in quality of life as measured by SF-36.
Groups:
- Afamelanotide: Subjects visited the clinic on Day 0 (administration of afamelanotide implant and porfimer sodium), Day 2 (photodynamic therapy), and Days 20 and 90 for assessments of adverse events, concomitant medication and the results of evaluation of phototoxicity.
  Afamelanotide
- Placebo: Subjects visited the clinic on Day 0 (administration of placebo implant and porfimer sodium), Day 2 (photodynamic therapy), and Days 20 and 90 for assessments of adverse events, concomitant medication and the results of evaluation of phototoxicity.
  Placebo
Arm/Group | Afamelanotide | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Quality of Life
Description: Quality of life, as measured by the Short Form-36 Health survey (SF-36) (quality of life questionnaire). The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Time Frame: From Day 0 to Day 20, Day 60 and Day 90
Measure: Mean (Full Range); unit: Scores on a scale
Arm/Group | Afamelanotide | Placebo
Number analyzed (Participants) | 7 | 5
Scores on a scale
  Day 20 - Day 0 (Physical functioning) | -5.7 [-35.0 to 0.00] | 8.0 [-15.0 to 30.0]
  Day 20 - Day 0 (Role Physical) | -14.6 [-56.3 to 6.3] | 0.0 [-18.8 to 50.0]
  Day 20 - Day 0 (Bodily Pain) | -1.4 [-28.0 to 78.0] | -11.6 [-68.0 to 59.0]
  Day 20 - Day 0 (General Health) | 2.0 [-25.0 to 60.0] | -27.6 [-43.0 to -13.0]
  Day 20 - Day 0 (Vitality) | -1.5 [-18.8 to 12.5] | -7.9 [-18.8 to 0.0]
  Day 20 - Day 0 (Social functioning) | 1.2 [-50.0 to 50.0] | 7.5 [-37.5 to 37.5]
  Day 20 - Day 0 (Role - Emotional) | -7.1 [-50.0 to 0.0] | 10.0 [-25.0 to 50.0]
  Day 20 - Day 0 (Mental Health) | 1.9 [-20.0 to 35.0] | 3.0 [-10.0 to 15.0]
  Day 20 - Day 0 (Physical Component Summary) | -2.6 [-13.1 to 2.7] | -4.8 [-18.4 to 10.6]
  Day 20 - Day 0 (Mental Component Summary) | 0.3 [-12.1 to 10.4] | 2.7 [-6.1 to 10.3]
  Day 60 - Day 0 (Physical Functioning) | -13.6 [-80.0 to 0.0] | -10.0 [-40.0 to 20]
  Day 60 - Day 0 (Role- Physical) | -8.9 [-56.3 to 12.5] | -13.8 [-43.8 to 31.3]
  Day 60 - Day 0 (Bodily Pain) | 2.0 [-28.0 to 52.0] | -21.4 [-68.0 to 19.0]
  Day 60 - Day 0 (General Health) | -4.2 [-32.0 to 18.0] | -33.0 [-47.0 to -20.0]
  Day 60 - Day 0 (Vitality) | 5.4 [-6.3 to 12.5] | -5.4 [-25.0 to 12.5]
  Day 60 - Day 0 (Social Functioning) | 0.0 [-50.0 to 37.5] | -17.5 [-50.0 to 25.0]
  Day 60 - Day 0 (Role- Emotional) | 6.0 [-50.0 to 91.7] | -10.0 [-50.0 to 25.0]
  Day 60 - Day 0 (Mental Health) | 2.9 [-10.0 to 10.0] | -2.0 [-20.0 to 10.0]
  Day 60 - Day 0 (Physical Component Summary) | -4.7 [-23.7 to 7.7] | -9.4 [-18.4 to 4.0]
  Day 60 - Day 0 (Mental Component Summary) | 4.3 [-8.6 to 34.2] | -2.5 [-17.6 to 4.8]
  Day 90 - Day 0 (Physical Functioning) | -13.6 [-80.0 to 5.0] | -5.0 [-40.0 to 30.0]
  Day 90 - Day 0 (Role- Physical) | 0.0 [-12.5 to 6.3] | -3.8 [-37.5 to 31.3]
  Day 90 - Day 0 (Bodily pain) | -2.7 [-16.0 to 19.0] | -13.8 [-69.0 to 19.0]
  Day 90 - Day 0 (General Health) | -4.1 [-27.0 to 15.0] | -32.0 [-60.0 to 13.0]
  Day 90 - Day 0 (Social Functioning) | 0.0 [-37.5 to 37.5] | -12.5 [-62.5 to 25.0]
  Day 90 - Day 0 (Role- Emotional) | 0.0 [-50.0 to 91.7] | -11.7 [-75.0 to 33.3]
  Day 90 - Day 0 (Mental Health) | -2.1 [-10.0 to 10.0] | -9.0 [-40.0 to 15.0]
  Day 90 - Day 0 (Physical Component Summary) | -3.0 [-23.7 to 8.2] | -5.1 [-14.7 to 6.4]
  Day 90 - Day 0 (Mental Component Summary) | 0.7 [-14.3 to 34.2] | -6.3 [-30.2 to 7.3]

ADVERSE EVENTS:
Description: None of the serious adverse events were deemed to be related to study drug
Arm/Group | Afamelanotide | Placebo
Serious Adverse Events (participants affected / at risk) | 2/9 | 3/7
Other Adverse Events (participants affected / at risk) | 6/9 | 1/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afamelanotide (N=9) | Placebo (N=7)
Haematemesis (Gastrointestinal disorders) | 0 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0
Overdose of Previscan (Fluindione) (Injury, poisoning and procedural complications) | 1 | 0
Drug toxicity (morphine) (Injury, poisoning and procedural complications) | 1 | 0
Subdiaphragmatic abscess (Infections and infestations) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afamelanotide (N=9) | Placebo (N=7)
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Headache (Nervous system disorders) | 3 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No